CLINICAL TRIAL: NCT03407521
Title: Measuring Response of Adding Isosorbide Mononitrate to Misoprostol in Induction of Second Trimester Abortion
Brief Title: Misoprosotol and Isosorbide Mononitrate for Induction of Second Trimester Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed abd elfatah elsenity, lecturer MD, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R02 MH12345
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Second Trimester Abortion
Keywords: second trimester abortion
MeSH Terms: interventions — Misoprostol; isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): misoprostol tab 200mcg 2 tab at first then one every 4 hours with isosorbide mononitrate 20mg once
  Interventions: Drug: Misoprostol; Drug: isosorbide mononitrate
- control group (Placebo Comparator): misoprostol tab 200mcg 2 tab at first then one every 4 hours with placebo
  Interventions: Drug: Misoprostol; Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — induction of abortion using misoprostol
Drug: isosorbide mononitrate — isosorbide mononitrate
  Arms: study group
Drug: Placebo — Placebo
  Arms: control group

SUMMARY:
the investigators aimed to study the efficacy and safety of nitric oxide donors when combined with prostaglandins in induction of second trimester abortion expecting that both drugs when used together will be of greater efficiency and associated with less side effects.

the study included 60 women with gestational age between 13weeks+0day and 26weeks+6days indicated for pregnancy termination due to maternal or fetal cause.

DETAILED DESCRIPTION:
the study aimed to compare the effect of isosorbid mononitrate when combined with misoprostol and misoprostol when used alone in second trimester abortion, expecting that both drugs when used together will be more effective and associated with fewer side effects.

In this study 60 women were enrolled, divided into two groups. The first group (group I), 30 women received misoprostol and isosorbid mononitrate.

The second group (group II), 30 women received misoprostol and placebo. The primary aim of the study was the occurrence of complete abortion in the first 24 hours.

The study concluded that the combination of isosorbid mononitrate with misoprostol is more effective in second trimester abortion than misoprostol with placebo, but is associated with more side effects mainly headache.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 -40 years
* Missed abortion
* Singelton pregnancy
* Gestationl age between 13 and 26 weeks of pregnancy
* Normal uterus and cevix on clinical examination
* Cervix is not dilatated
* No uterine activity and vaginal bleeding
* Written and informed consent by the patient
* Unscarred uterus

Exclusion Criteria:

* Presence of uterine contraction or bleeding
* Evidences suggesting of onset of spontaneous abortion as Previous trial to induce abortion
* Multifetal pregnancy
* Suspicion of septic abortion
* History of cervical surgery or manipulation
* Uterine anomaly
* IUD in situ
* Associtaed hemorrhagic disorder
* History of adverse effects to vaginally adminstered medication
* Inability to insert vaginal medication high in vagina

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
induction abortion interval | 24 hours
  time needed to induce abortion in second trimester abortion

CONTACTS AND LOCATIONS:
Overall Officials: mohamed ab elsenity, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
publish in scientific journals

REFERENCES:
- [Result] Jain JK, Mishell DR Jr. A comparison of misoprostol with and without laminaria tents for induction of second-trimester abortion. Am J Obstet Gynecol. 1996 Jul;175(1):173-7. doi: 10.1016/s0002-9378(96)70270-3. PMID 8694046